CLINICAL TRIAL: NCT05250479
Title: Effect of Mindfulness Education on Fear of Childbirth, Mode of Delivery, Childbirth Experience and Prenatal and Maternal Attachment in Primiparous Pregnant Women
Brief Title: Effect of Mindfulness Education in Primiparous Pregnant Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, Özlem AKIN, Lecturer, PhD student, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: ozlem20
Record Dates: First submitted 2022-01-30; First posted 2022-02-22 (Actual); Last update posted 2022-02-22 (Actual); Status verified 2022-02

CONDITIONS: Pregnancy Related; Mindfulness; Fear of Childbirth; Attitude
Keywords: primiparous; pregnant women; fear of childbirth; prenatal attachment; mindfulness education; childbirth experiences; mode of birth; maternal attachment; nursing
MeSH Terms: conditions — Behavior

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 44 pregnant women won't receive mindfulness training
- experimental group "mindfulness education" (Experimental): mindfulness education 44 pregnant women will receive mindfulness training
  Interventions: Behavioral: Mindfulness education

INTERVENTIONS:
Behavioral: Mindfulness education — 44 primiparous pregnant women will receive mindfulness education
  Arms: experimental group "mindfulness education"

SUMMARY:
While adaptation is generally achieved to the psychological changes that develop during pregnancy, some women may experience psychological changes such as contradiction, uncertainty, introversion, passive personality, addiction, fear, and anxiety in different periods of pregnancy. During this period, the fear of childbirth may also be experienced in pregnant women. Fear of childbirth or tokophobia is a phobic condition in which a woman avoids giving birth despite desperately wanting a baby. While fear of childbirth can have a negative impact on women's psychological health during pregnancy and birth experience, it is associated with negative obstetric outcomes and postpartum mental health problems. It is possible that the fear of childbirth reduces the mother's attachment to the fetus. Fear increases avoidant attachment and anxiety, which may be associated with lower commitment scores. There is a strong relationship between fear of childbirth and negative birth outcomes. Both affect the psychological well-being of the mother, adjustment to motherhood, and the quality of the mother's relationship with the baby. Knowing the fear of childbirth is important as it is associated with various health problems such as certain physiological and obstetric disorders and they can increase the possibility of emergency cesarean section. Mindfulness-based interventions combine elements of established cognitive behavioral therapy and psychoeducational content to support a self-effective approach to reduce stress-related symptoms and improve mental and physical well-being. Mindfulness-based practices that involve focusing on the present moment and accepting life without judgment are one of the effective ways to prepare for childbirth, help women feel more empowered and aware of their motherhood processes, and give mothers the opportunity to share knowledge and emotions. Mindfulness-based birth education intervention appears to be applicable for women and is associated with improvements in women's sense of control and confidence in giving birth.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years
* 28-32. in gestational week
* First pregnancy
* Understands and speaks Turkish
* Single pregnancy
* Having at least primary school education

Exclusion Criteria:

* Having a high-risk pregnancy
* Receiving psychotherapy or medication in the last six months before the study
* with chronic disease Participating in childbirth preparation courses Planning a cesarean delivery with a diagnosed psychiatric illness Pregnant women with previous yoga and meditation experience Pregnant women with a high gestational age will be excluded from the study due to the possibility of giving birth before the end of the follow-up period

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Enrollment: 88 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2022-12-20 (Estimated); Study Completion 2023-06-20 (Estimated)

PRIMARY OUTCOMES:
Wijma Delivery Expectancy/Experience Questionnaire A (W-DEQ A) | 28-32. pregnant women
  determining the level fear of childbirth
Wijma Delivery Expectancy/Experience Questionnaire A (W-DEQ A) | After 32 weeks of pregnancy
  determining the level fear of childbirth
Prenatal Attachment Inventory | 28-32. pregnant women
  determine prenatal mother-infant attachment
Prenatal Attachment Inventory | After 32 weeks of pregnancy
  determine prenatal mother-infant attachment

SECONDARY OUTCOMES:
Maternal Fetal Attachment Scale | postpartum 1st month
  determine maternal fetal attachment
Wijma Delivery Expectancy/Experience Questionnaire B (W-DEQ B) | postpartum 1st month
  determining the level fear of childbirth

CONTACTS AND LOCATIONS:
Overall Officials: Nülüfer Erbil, PhD, Study Director — Ordu University
Locations (1):
- Recep Tayyip Erdogan University Training and Research Hospital, Rize, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No